CLINICAL TRIAL: NCT06021457
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of RBT-1 on Reducing the Risk of Post-Operative Complications in Subjects Undergoing Cardiac Surgery
Brief Title: Effect of RBT-1 on Reducing the Risk of Post-Operative Complications in Subjects Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REN-007
Record Dates: First submitted 2023-08-17; First posted 2023-09-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Post-Operative Complications in Cardiac Surgery
Keywords: Cardiac Surgery; CABG; Valve; Cardiopulmonary Bypass; Preconditioning

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to RBT-1 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RBT-1 (Experimental): Single IV infusion prior to cardiac surgery
  Interventions: Drug: RBT-1
- Placebo (Placebo Comparator): Single IV infusion prior to cardiac surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBT-1 — Intravenous administration
  Arms: RBT-1
Drug: Placebo — Intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of RBT-1 on reducing the risk of post-operative complications in subjects undergoing cardiac surgery on cardiopulmonary bypass (CPB). A sub-study will also be conducted to evaluate the pharmacokinetic (PK) profile of a single administration of RBT-1 by means of a popPK approach in subjects scheduled to undergo cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at Screening.
2. Planned to undergo non-emergent CABG and/or cardiac valve surgery requiring CPB; non-emergent surgery must allow for study drug infusion ≥24 but ≤48 hours prior to surgery.
3. If female, subjects must use an effective method of birth control or abstain from sexual relations with a male partner (unless has undergone tubal ligation or hysterectomy or is at least 1 year postmenopausal) for the duration of their study participation.
4. If male, subjects must use an effective method of birth control or abstain from sexual relations with a female partner for the duration of their study participation, unless the subject has had a vasectomy ≥6 months prior to infusion with study drug.
5. Willingness to comply with all study-related procedures and assessments.

Exclusion Criteria:

1. Surgery planned to occur <24 hours from the start of study drug infusion.
2. Presence of acute organ dysfunction (AKI, acute decompensated heart failure, acute respiratory failure, stroke, etc) as assessed by the Investigator at the time of Screening.
3. Surgery to be performed without CPB.
4. Chronic kidney disease (CKD) requiring dialysis.
5. Hypokalemia and/or hypomagnesemia within 24 hours prior to study drug infusion; electrolytes can be replenished if low.
6. Cardiogenic shock or immediate requirement for inotropes, vasopressors, or other mechanical devices, such as intra-aortic balloon pump (IABP).
7. Known history of cancer within the past 2 years, except for carcinoma in situ of the cervix or breast, early-stage prostate cancer, or adequately treated non-melanoma cancer of the skin.
8. Known or suspected sepsis at time of Screening.
9. Asplenia (anatomic or functional).
10. History of hemochromatosis, iron overload, or porphyria.
11. Known hypersensitivity or previous anaphylaxis to SnPP or FeS.
12. Female subject who is pregnant or breastfeeding.
13. Participation in a study involving an investigational drug or device within 30 days prior to study drug infusion or throughout participation in REN-007.
14. In the opinion of the Investigator, for any reason, the subject is an unsuitable candidate to receive RBT-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite of the following outcomes: death, incidence of AKI requiring dialysis, 30-day cardiopulmonary readmission, and intensive care unit (ICU days). | Index hospitalization (ie, hospitalization post-cardiac surgery up to 60 days) or within 30-days post-discharge, as applicable
  The analysis will be based on a "win ratio," which uses the Finkelstein-Schoenfeld method wherein all RBT-1 patients are paired with all placebo patients; each pair is declared to be a win for RBT-1, a win for placebo, or a tie, based on the hierarchical composite. The win ratio is the ratio of the number of wins for RBT-1 divided by the number of wins for placebo.

SECONDARY OUTCOMES:
Composite of the Number of Post-operative Complications | Index hospitalization (ie, hospitalization post-cardiac surgery up to 60 days) or within 30-days post-discharge, as applicable
  The number of the following post-operative complications per patient will be assessed:
  * Death
  * AKI requiring dialysis
  * >3 days in ICU
  * >24 hours on ventilator
  * 30-day cardiopulmonary readmission
  * Need for blood transfusion during index hospitalization
  * New-onset atrial fibrillation during index hospitalization
ICU Days | Index hospitalization (ie, hospitalization post-cardiac surgery up to 60 days)
  Days in ICU
30-day Cardiopulmonary Readmission Rates | Within 30-days post-discharge
  Readmissions due to cardiopulmonary reasons

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — World Health Research Institute
Locations (37):
- United States (30):
  - Research Site, Huntsville, Alabama
  - Research Site, La Jolla, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Flushing, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
- Canada (7):
  - Research Site, Kelowna, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No